CLINICAL TRIAL: NCT02138760
Title: Comparison of MRI Fusion Biopsy Techniques in Men With Elevated PSA and Prior Negative Prostate Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, David S Finley, MD, Director of Robotic Surgery, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KP-MRI-2014
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate biopsy; magnetic resonance imaging guidance; detection rates; performance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI guided cognitive fusion biopsy (No Intervention): Men in this arm will undergo MRI followed by systematic biopsy and then additional cognitive (freehand) biopsies of MRI suspicious targets
- UroNav fusion biopsy (Experimental): Men in this arm will undergo MRI followed by systematic biopsy and then additional UroNav fusion biopsy of MRI suspicious targets
  Interventions: Procedure: MRI UroNav fusion biopsy

INTERVENTIONS:
Procedure: MRI UroNav fusion biopsy
  Other Names: UroNav (InVivo corp)
  Arms: UroNav fusion biopsy

SUMMARY:
Men with elevated prostate specific antigen bloodtest and prior negative prostate biopsy have a 30-60% of harboring occult prostate cancer. Multiparametric magnetic resonance imaging (mpMRI) is an imaging test that may improve prostate cancer detection rates in this population of men. In this prospective randomized trial multicenter trial the investigators will assess the detection rates of prostate cancer diagnosis of systematic biopsy compared with the addition of either a computer targeted system (UroNav - InVivo corp) to sample suspicious areas identified on mpMRI versus the detection rate mpMRI guided freehand biopsy (cognitive fusion biopsy). The hypothesis being tested is that computerized fusion guided biopsy (UroNav) will increase detection prostate cancer compared to cognitive biopsy of these areas and systematic biopsy alone.

DETAILED DESCRIPTION:
Prostate cancer (PC) is the second most common cancer in men in the United States, affecting approximately 250,000 men per year. With the advent of the prostate specific antigen (PSA) blood test, PC has undergone downward stage migration resulting in earlier cancer detection. In the pre-PSA era, tumors presented with advanced stage which were often visible on transrectal ultrasound. In the modern era, tumors more often are microscopic and not apparent on ultrasound imaging which creates a diagnostic challenge in which biopsy is essentially blind. As a result, many tumors are missed resulting in subsequent biopsies, tumor progression, and decreased cancer-specific survival due to delayed diagnosis.

Multiparametric magnetic resonance imaging (mpMRI) of the prostate has now become the preferred imaging modality to visualize prostate tumors radiographically. mpMRI has become increasing utilized for targeting tumor suspicious areas in the prostate in men with prior negative conventional systematic biopsy. Numerous studies have shown MRI targeted biopsy results in detection of cancer in this subset of men in approximately 30-60% of patients (refs). In addition, MRI detects a higher number of aggressive prostate cancers which would require treatment.

Several methods of incorporating MRI into biopsy targeting have been tested: 1) in gantry/in bore MRI biopsy 2) Robotic biopsy (Artemis) 3) UroNav ultrasound-MR fusion biopsy. The first two techniques are cumbersome and difficult to use in clinical practice. The latter technology is the most widely utilized, user and patient friendly technique. UroNav utilizes a work-station which imports the MRI and then co-registers (fuses) it with real time ultrasound; the ultrasound transducer communicates with an electromagnetic received above the patient to allow the work-station/computer to target suspicious MRI lesions to guide the users needle to the appropriate 3-dimensional location. Data has shown this to be more effective than either systematic biopsy or free-MRI guided biopsy.

The goal of the present study is to compare head-to-head systematic biopsy + freehand MRI targeted biopsy vs systematic biopsy + UroNav targeted in men with elevated PSA and prior negative systematic biopsy.

ELIGIBILITY:
Inclusion Criteria:

* PSA > 2.5 ng/ml (ages 30-50) or PSA > 4.0 ages (50-79)
* Patients with prior negative prostate biopsy
* Written informed consent
* Age > 30

Exclusion Criteria:

* Prior diagnosis of prostate cancer
* Age> 79
* No contraindication to MRI or prostate biopsy (e.g. coagulopathy, severe medical comorbidity prohibiting halting of anticoagulation therapies, anatomical contraindications)
* Active urinary tract infection or indwelling catheter
* Prior pelvic irradiation
* Prior androgen deprivation hormonal therapy
* Prostate surgery (e.g. prostate biopsy, transurethral prostate procedure) within 8 weeks prior to mpMRI.
* Contraindication to MRI (extreme claustrophobia, metallic implants incompatible with MRI)

Ages: 30 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer detection rate | 1 week after biopsy
  Prostate cancer detection rate between MRI guided free hand biopsy and UroNav targeted biopsy

SECONDARY OUTCOMES:
Clinically significant prostate cancer detection rate | 1 week after biopsy
  Detection rate between techiques of Gleason 4 or higher prostate cancer

OTHER OUTCOMES:
Tumor volume | 1 week after biopsy
  % core involvement of cancer between techniques

CONTACTS AND LOCATIONS:
Overall Officials: David S Finley, MD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente Los Angeles (Sunset), Los Angeles, California
  - Kaiser Permanente Riverside, Riverside, California